CLINICAL TRIAL: NCT01079832
Title: A Prospective Evaluation of a Palliative Radio-Surgical Approach for the Treatment of Gynecologic Malignancies
Brief Title: Stereotactic Radiosurgery Using CyberKnife in Treating Women With Advanced or Recurrent Gynecological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE13808; NCI-2010-00285 (Other: NCI/CTRP); CASE13808 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Fallopian Tube Cancer; Ovarian Sarcoma; Ovarian Stromal Cancer; Recurrent Cervical Cancer; Recurrent Endometrial Carcinoma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Uterine Sarcoma; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer; Stage III Cervical Cancer; Stage III Endometrial Carcinoma; Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage III Uterine Sarcoma; Stage III Vaginal Cancer; Stage III Vulvar Cancer; Stage IV Endometrial Carcinoma; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Uterine Sarcoma; Stage IV Vulvar Cancer; Stage IVA Cervical Cancer; Stage IVA Vaginal Cancer; Stage IVB Cervical Cancer; Stage IVB Vaginal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I: CyberKnife Radiosurgery (Experimental): Patients undergo 3 fractions of CyberKnife stereotactic radiosurgery.
  Interventions: Radiation: stereotactic radiosurgery; Procedure: quality-of-life assessment

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Radiation will be delivered in 3 fractions. The dose level will range between 500 to 800cGy per fraction at the discretion of the treating radiation oncologist
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: Stereotactic radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This clinical trial studies stereotactic radiosurgery using CyberKnife works in treating women with advanced or recurrent gynecological malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary goal of this study is to estimate the rate of grade 3 or higher acute toxicities observed during a 6 month period following CyberKnife radiosurgery for gynecologic cancers.

II. To evaluate clinical response to radio-surgery for gynecologic tumors.

III. To assess general and site specific quality of life (using SF-12, FACT-En, FACT-O, FACT-Cx or FACT-V) and to evaluate patient's level of pain.

SECONDARY OBJECTIVES:

I. As a secondary objective, toxicities during the 2 years following CyberKnife radiosurgery will also be described.

OUTLINE:

Patients undergo 3 fractions of CyberKnife stereotactic radiosurgery.

After completion of study treatment, patients are followed at 1, 3, 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion

* Pathologically proven gynecologic malignancy
* No prior cryosurgery or radiofrequency ablation, in target lesion
* Patient is able to give and sign study specific informed consent
* Measurable disease, according to RECIST criteria
* Laboratory parameters and appropriate clearance from anesthesia based on other medical co-morbidities for placement of fiducials; these would include CBC, basic metabolic panel, BUN, and creatinine
* >= 4 weeks from previous treatment (chemotherapy or radiation) of malignancy
* ECOG performance status of 0-3 as this procedure is minimally invasive and considered palliative in these patients

Exclusion

* Any patient with active connective tissue disease such as lupus or dermatomyositis is excluded
* Any patient with active Crohn's disease or active ulcerative colitis is excluded
* Major medical or psychiatric illness, which would prevent completion of treatment or interfere with follow-up is excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert DeBernardo, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 24,2009 and September 7, 2011, 50 patients were recruited from University Hospitals in Cleveland Ohio.
Period: Overall Study
Arm/Group | Arm I: CyberKnife Radiosurgery
Started | 50
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I: CyberKnife Radiosurgery
Number analyzed (Participants) | 50
Age Continuous [Median (Full Range); unit: years] | 66 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Acute Toxicity Rate
Description: The incidence of grade 3 or 4 possible SBRT-related non-hematological toxicities observed during a 6 month period.
Time Frame: at 6 months after treatment
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: CyberKnife Radiosurgery
Number analyzed (Participants) | 50
percentage of participants | 6

2. Secondary Outcome: Disease-free Survival
Description: Median disease free survival
Time Frame: completion of study at 24 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: CyberKnife Radiosurgery
Number analyzed (Participants) | 50
months | 7.8 [4 to 11.6]

3. Secondary Outcome: Median Overall Survival
Description: Length of time patients survived at study end.
Time Frame: 24 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: CyberKnife Radiosurgery
Number analyzed (Participants) | 50
months | 20.2 [10 to 29.5]

4. Secondary Outcome: Quality of Life
Time Frame: After completion of study treatment, patients are followed at 1, 3, 6, 12, 18 and 24 months.
Population: Participant surveys were unreliably returned to investigators, making this analysis not meaningful.
Arm/Group | Arm I: CyberKnife Radiosurgery
Number analyzed (Participants) | 0

5. Secondary Outcome: Clinical Response Rate
Description: Percentage of patients with a clinical response following RECIST (Response Evaluation Criteria in Solid Tumors) Criteria: Confirmed complete response(CR), Stable disease (SD), partial response (PR), or without progressive disease (PD).
Time Frame: at 6 months from study entry
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: CyberKnife Radiosurgery
Number analyzed (Participants) | 50
percentage of participants | 68 [53 to 80]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while patients were receiving treatment and during 6 months of follow up.
Arm/Group | Arm I: CyberKnife Radiosurgery
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 34/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: CyberKnife Radiosurgery (N=50)
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1 — Additional adverse events associated with this hospitalization were: Grade 1 INR (International Normalized Ratio of prothrombin time) Grade 2 Liver dysfunction/failure (clinical)
Confusion (Nervous system disorders) | 1 — Confusion - Brain metastasis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Arm I: CyberKnife Radiosurgery (N=50)
Hemoglobin (Blood and lymphatic system disorders) | 6/34
Platelets (Blood and lymphatic system disorders) | 3/34
"Fatigue (asthenia, lethargy, malaise)" (General disorders) | 10/34
Anorexia (Metabolism and nutrition disorders) | 2/34
Diarrhea (Gastrointestinal disorders) | 3/34
Nausea (Gastrointestinal disorders) | 6/34
Pain - Abdomen NOS (Gastrointestinal disorders) | 2/34
Edema: limb (General disorders) | 2/34
Creatinine (Metabolism and nutrition disorders) | 2/34
Pain - Back (Musculoskeletal and connective tissue disorders) | 3/34
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 2/34
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes